CLINICAL TRIAL: NCT05505058
Title: One-time Informed Consent for Research in Prison: A Randomized Comparison Between Audio-visual and Written Materials
Brief Title: One-time Informed Consent for Research in Prison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Stéphanie Baggio, PD Dr., University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-01797
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Informed Consent
Keywords: Prison; Research ethics; Audio-visual intervention; Bioethics; Human rights

STUDY DESIGN:
Intervention Model Description: Cross-sectional study with parallel randomized design (allocation 1:1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audio-visual material (Experimental): The video for informed consent was developed by a science filmmaker (https://www.lostlikebeesinrain.comhttps://betomation.space/) for the project's purposes.
  Interventions: Behavioral: Audio-visual material
- Paper-based conventional material (Active Comparator): The written material for informed consent was developed by the Swiss Association of Research Ethic Committees and the booklet was designed by the Clinical Research Center of the Geneva University Hospitals.
  Interventions: Behavioral: Audio-visual material

INTERVENTIONS:
Behavioral: Audio-visual material — Participants were randomized to receive a paper-based conventional material or to watch a 4-min video. Materials both included legal information required by the Swiss Federal Act on Research involving Human Beings.
  Other Names: Paper-based conventional material

SUMMARY:
Ethical research on detained persons remains limited, including research on informed consent. This study aimed to fill in this research gap and compared audio-visual and paper-based materials for a one-time general informed consent for research in prison, using a randomized design. The primary outcome was whether participants sign the inform consent. Secondary outcomes included understanding, evaluation, and time to read/watch the informed consent.

DETAILED DESCRIPTION:
Detained persons constitute a very vulnerable and perhaps reluctant to share their medical data. In particular, it is crucial to ensure that these persons, deprived of their liberty, understand that their consent is voluntary and that a refusal will not have any consequence on their treatment or care. In other words, it is necessary to ensure that consent is informed. In a historical context of non-ethical research using detained persons, this is a crucial issue. However, while detained persons are now protected from various forms of abuse, this may have had the consequence of reducing research involving them, to the detriment of understanding their characteristics and vulnerabilities.

A general consent for research will encourage research on prison populations by facilitating access to their medical data in order to study and reduce health disparities, for this population with multiple somatic and psychiatric comorbidities.

Our main questions are:

Q1. What is the acceptability rate of general consent for research in detained persons? Q2. What are the characteristics (socio-demographic and medical) of detained person who refuse to give their consent? Q3. Which material (paper-based or video) is more effective?

To answer these research question, we will use an exploratory randomized cross-sectional trial, conducted in an adult pre-trial prison and a juvenile detention center. Participants will be randomly assigned to read or watch information about informed consent, stratified on the prison. In both prisons, the study will take place in the prison medical unit.

This project is aimed to improve general consent, which contributes to reducing inequalities in documentation on health status, and ultimately, health inequalities.

ELIGIBILITY:
Inclusion Criteria:

* to be18 years old or more in the adult prison and 14 years old or more in the juvenile detention center
* to be able to communicate in one of the languages of the study material
* to agree to participate in this study.

Exclusion Criteria:

* presence of an acute psychiatric problem preventing the person from participating in the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptance to sign the informed consent | Assessed immediately after intervention
  Binary outcome, legal Swiss document

SECONDARY OUTCOMES:
Understanding of the informed consent | Assessed immediately after intervention
  Eight self-developed questions assessed as true/false and combined in a 0-8 points score
Evaluation of the informed consent | Assessed immediately after intervention
  Nine self-developed question assessed on a six-point Likert scale and averaged
Time to read/watch | Assessed immediately after intervention
  Time in minutes for reading the booklet (the video has a unique duration of 4 min)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Wolff, MD, Study Chair — Division of Prison Health, Geneva University Hospitals
Locations (1):
- Division of prison health, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
The datasets are not publicly available due their sensitive nature (detained persons) but are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Baggio S, Getaz L, Giraudier L, Tirode L, Urrutxi M, Carboni S, Britan A, Price RL, Wolff H, Heller P. Comparison of Audiovisual and Paper-Based Materials for 1-Time Informed Consent for Research in Prison: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2235888. doi: 10.1001/jamanetworkopen.2022.35888. PMID 36219446